CLINICAL TRIAL: NCT04838405
Title: A Phase 1 Randomized, Double Blind, Placebo Controlled, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CT-388 in Otherwise Healthy Overweight and Obese Adult Participants and in Obese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of CT-388 in Otherwise Healthy Overweight and Obese Adults and Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carmot Therapeutics, Inc. (Industry)
Collaborators: Carmot Australia First Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-388-101
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CT-388 (Experimental): SC dose of CT-388
  Interventions: Drug: CT-388
- Placebo (Placebo Comparator): SC dose of placebo matching CT-388 dose
  Interventions: Drug: Placebo
- CT-388 Optional (Experimental): SC dose of CT-388
  Interventions: Drug: CT-388
- CT-388 MD (Experimental): SC dose of CT-388
  Interventions: Drug: CT-388

INTERVENTIONS:
Drug: CT-388 — Synthetic Peptide
  Arms: CT-388; CT-388 MD; CT-388 Optional
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a first-in-human evaluation of CT-388 in a double blind, placebo controlled, randomized, SAD/MAD/MD, safety, tolerance, PK, and PD study when administered as a SC injection in otherwise healthy overweight and obese adult participants and obese participants with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Males or females
* 18-65 years old, inclusive
* BMI 27.0-40.0, inclusive
* Stable body weight for 2 months

Exclusion Criteria:

* Significant medical history
* Uncontrolled hypertension
* History of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by self-report | Baseline up to 24 weeks
  Safety and tolerability

SECONDARY OUTCOMES:
Area under the concentration versus time curve (AUC) | Baseline up to 24 weeks
  PK AUC
Maximum observed drug concentration (Cmax) | Baseline up to 24 weeks
  PK Cmax
Elimination half-life | Baseline up to 24 weeks
  PK t1/2
Change in mean body weight | Baseline up to 24 weeks
  PD body weight
Change in mean glucose levels | Baseline up to 24 weeks
  PD glucose
Change in mean insulin levels | Baseline up to 24 weeks
  PD insulin

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Carmot Therapeutics, Inc.
Locations (2):
- Carmot Clinical Research Unit 101, Perth, Western Australia, Australia
- Carmot Clinical Research Unit 105, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Carmot Therapeutics, Inc. — https://carmot-therapeutics.us/